CLINICAL TRIAL: NCT03169673
Title: Healthy Lung Study- Development of 3 Tesla MRI Hardware and Software for Helium-3 Gas Imaging of the Lung: Healthy Volunteer Development Study
Brief Title: Healthy Lung Study- Development of 3T MRI Hardware and Software for 3He Gas Imaging of the Lung: Healthy Volunteer Development Study
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Other Study IDs: ROB0006
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers
Keywords: Magnetic Resonance Imaging; Pulmonary Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Hyperpolarized Helium 3 Magnetic Resonance Imaging — Hyperpolarized noble gas imaging using Helium-3 has been used to explore structural and functional relationships in the lung in patients with lung disease and healthy controls. In contrast to proton-based MRI imaging, 3He gas is used as a contrast agent to directly visualize the airways, and thus ventilation. Whereas the normal density of gas is too low to produce an easily detectable signal, this is overcome by artificially increasing the amount of polarization per unit volume using optical pumping.

SUMMARY:
Healthy volunteers aged 18-75 will undergo hyperpolarized 3-Helium MRI and pulmonary function testing for the development of tools to assess image signal to noise and reproducibility of spin-density and diffusion-weighted imaging.

DETAILED DESCRIPTION:
During a two hour visit, subjects will provide written informed consent and then undergo: 1) brief medical history and vital signs, 2) full pulmonary function tests, 3) proton MRI, 4) spin-density and/or diffusion weighted 3He MRI.

Full pulmonary function tests including spirometry, plethysmography and diffusing capacity of carbon monoxide (DLCO), Lung Clearance Index (LCI) and Airwave Oscillometry (AO) will be performed according to ATS guidelines. MedGraphics Elite Series, MedGraphics Corporation. St. Paul, MN USA and/or nDD EasyOne Spirometer, nDD Medical Technologies Inc. Andover, MA USA will be used. All measurements will be performed in the Pulmonary Function Laboratory at Robarts Research Institute.

Subjects will be placed in the 3T MR scanner with the 3He chest coil fitted over their torso and chest. Hearing protection will be provided to each subject to muffle the noise produced by the gradient RF coils. A pulse oximeter lead will be attached to all of the subjects to monitor their heart rate and oxygen saturation. MRI will be performed for up to a period of 30 minutes. All subjects will have supplemental oxygen available via nasal cannula at a flow-rate of 2 liters per minute as a precaution in the event of oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform a breath hold for up to 16 seconds.
* BMI between 18 and 40.
* Stable health on the basis of medical history.
* Smoking history < 1 pack/year.

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material.
* Subject has a daytime room air oxygen saturation <90% while lying supine.
* Patient is unable to perform spirometry or plethysmography maneuvers
* Patient is pregnant
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2007-09-21 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Ventilation Defect Percent (VDP) | 5 years
  VDP is a widely used noble gas MRI biomarkers that is calculated by normalizing ventilation defect volume to the thoracic cavity.

SECONDARY OUTCOMES:
Apparent Diffusion Coefficients (ADC) | 5 years
  Diffusion weighted noble gas MRI provides a way to quantify pulmonary microstructure by sensing the movements of inhaled gas atoms. The "apparent" dif fusion coefficient (ADC) during the diffusion time interval can be used to reflect the extent of alveolar restriction of gas atom movements, providing a surrogate measurement of airspace dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Study Principal Investigator Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capaldi DPI, Guo F, Xing L, Parraga G. Pulmonary Ventilation Maps Generated with Free-breathing Proton MRI and a Deep Convolutional Neural Network. Radiology. 2021 Feb;298(2):427-438. doi: 10.1148/radiol.2020202861. Epub 2020 Dec 8. PMID 33289613